CLINICAL TRIAL: NCT06400563
Title: Evaluation of the Magnetic Resonance-guided (MRg) Near-infrared Spectroscopy (NIRS) Imaging System Platform in Breast Cancer Patients
Brief Title: MRg-NIRS Imaging System Breast Cancer Trial
Acronym: MRg-NIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keith D. Paulsen (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Sponsor-Investigator, Keith D. Paulsen, Professor of Engineering, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY02001582
Record Dates: First submitted 2024-04-11; First posted 2024-05-06 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: MRI; MRg-NIRS; Near-infrared Spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study team will collect MRI-derived region of interest (ROI) data with T1, T2 and DCE-MRI sequences from 20 women with breast abnormalities and NIRS data concurrently. The study team will test whether the breast interface can provide optical measurements with positional data sensitivity >1%.
  The study team will conduct two interim analyses of optical sensitivity after completion of 5-10 patient exams to decide whether the breast interface should be modified.
  The breast interface is a non-significant risk device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MR-guided NIRS (Other): The MRg-NIRS device will be tested to see if it accommodates different breast sizes, covers the breast fully, includes the axilla, is compatible with commercial breast MRI coil and/or biopsy systems, and the signal-to-noise ratio is high enough for MRg-NIRS image reconstruction.
  The study team will collect MRI-derived ROI data with T1, T2 and DCE-MRI sequences from 20 women with breast abnormalities and NIRS data concurrently. The study team will also collect diffuse optical signals at 48x48 detector source positions over one side of breast at 6 wavelengths.
  Interventions: Device: MRg-NIRS

INTERVENTIONS:
Device: MRg-NIRS — The trial tests the investigator designed and developed Magnetic Resonance-guided (MRg) Near-infrared Spectroscopy (NIRS) imaging system for breast cancer detection. The wearable NIRS imaging system uses 8 flex circuit strips, each with six photo-detectors (PDs) and six source fibers, that are ready to attach to a breast radially by using an adhesive nipple cover and breast tape.
  Other Names: MR-guided NIRS Data Collection

SUMMARY:
This trial is a study of 20 women with breast cancer to evaluate the addition of MR-guided (MRg) near-infrared spectroscopy (NIRS) with and without contrast, as part of a program to improve clinical management of women receiving breast magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
This trial is designed to determine if the MRg-NIRS system will contribute significantly to improved clinical management of women receiving breast magnetic resonance imaging (MRI) by achieving diagnostic performance comparable to or better than dynamic contrast-enhanced (DCE) breast MRI alone.

The purpose of this clinical trial is to evaluate the addition of MRg-NIRS with and without contrast in 20 women with breast cancer. The women enrolled in the trial will be those who have a newly diagnosed breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females age ≥ 18 years old
2. Participants capable of providing written informed consent
3. Women with a recent diagnosis of breast cancer.
4. Women who are in pre-surgical planning must have an estimated tumor size of 2.0 cm or less on available imaging.
5. Women who are in pre-surgical planning must have had a breast biopsy at least 10 days prior to the MRg-NIRS exam.

Exclusion Criteria:

1. Participants with absolute or relative contraindication to MRI:

   1. the presence of an electronic implant, such as a pacemaker
   2. the presence of a metal implant, such as an aneurysm clip
   3. claustrophobia
   4. renal failure (FDA's guidance for gadolinium of a creatinine clearance less than 30 mL/1.73 m2 BSA)
2. Pregnant women
3. Breast implants
4. Prisoners
5. Participants with visually inadequate healing from breast biopsy.

Ages: 18 Years to 83 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Optical sensitivity of the MRg-NIRS platform | up to one hour on day of MRI
  Optical data sensitivity will be measured (The sensitivity of the measurements to a given region identified by MRI, Sr, will be calculated as the sum of the log of the Jacobian times vector r. Here, r is a logical vector that identifies points within the region of interest and J is the Jacobian, the rate of change of measurements to a change in optical properties at a location in the region identified).

SECONDARY OUTCOMES:
Diagnostic performance of the MRg-NIRS platform | up to one hour on day of MRI
  Diagnostic performance will be measured in terms of sensitivity, specificity and area under the receiver-operator characteristic curve (ROC).

CONTACTS AND LOCATIONS:
Overall Officials: Keith D. Paulsen, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No